CLINICAL TRIAL: NCT02897765
Title: An Open-label, Phase IB Study of NEO-PV-01 + Adjuvant With Nivolumab in Patients With Melanoma, Non-Small Cell Lung Carcinoma or Transitional Cell Carcinoma of the Bladder
Brief Title: A Personal Cancer Vaccine (NEO-PV-01) w/ Nivolumab for Patients With Melanoma, Lung Cancer or Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech US Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: BioNTech SE (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-001
Record Dates: First submitted 2016-08-12; First posted 2016-09-13 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Urinary Bladder Cancer; Bladder Tumors; Transitional Cell Carcinoma of the Bladder; Malignant Melanoma; Melanoma; Skin Cancer; Carcinoma, Non-Small-Cell Lung; Lung Cancer
Keywords: Checkpoint Inhibitor; Immunotherapy; Personal Vaccine; Neoantigen; Poly-ICLC; Peptide
MeSH Terms: conditions — Urinary Bladder Neoplasms; Melanoma; Skin Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Nivolumab; Adjuvants, Pharmaceutic; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug: NEO-PV-01 + Nivolumab + Adjuvant (Experimental): Nivolumab at a dose of 240 mg administered by intravenous (IV) infusion over 30 minutes every two weeks. At Week 12, all patients, regardless of their disease status, will receive NEO-PV-01 + adjuvant administered subcutaneously (one vial of pooled peptides per injection site) in up to four distinct sites (each extremity or flanks) while continuing therapy with nivolumab.
  Interventions: Biological: NEO-PV-01; Biological: Nivolumab; Other: Adjuvant

INTERVENTIONS:
Biological: NEO-PV-01 — Personal cancer vaccine
  Other Names: Personal cancer vaccine
Biological: Nivolumab — monoclonal antibody against PD1
  Other Names: Opdivo
Other: Adjuvant — immune adjuvant
  Other Names: Hiltonol; poly-ICLC

SUMMARY:
The purpose of this study is to evaluate if the treatment with NEO-PV-01 + adjuvant in combination with nivolumab is safe and useful for patients with certain types of cancer. The study also will investigate if NEO-PV-01 + adjuvant with nivolumab may represent a substantial improvement over other available therapies such as nivolumab alone. All eligible patients will receive NEO-PV-01 + adjuvant and nivolumab while on this trial.

DETAILED DESCRIPTION:
This clinical trial will enroll patients with metastatic or advanced melanoma, lung, or bladder cancer. The three agents being used in this study are:

* A new, investigational, personal cancer vaccine called "NEO-PV-01"
* Poly-ICLC (Hiltonol), an investigational adjuvant that is used to help stimulate the immune system
* A cancer drug called nivolumab (OPDIVO®)

These agents are considered immunotherapy and work by stimulating the immune system to fight cancer. NEO-PV-01 is a truly personal vaccine therapy in that it is custom designed and manufactured to include targets for the immune system that are present uniquely on an individual's cancer. Poly-ICLC is an adjuvant that helps stimulate the immune system and make the vaccine, NEO-PV-01 more effective. Nivolumab helps T-cells, a certain type of immune cell, that recognize these targets to reach and attack the tumor. Nivolumab is in clinical development for treatment of bladder cancer and is approved by the FDA (the U.S. Food and Drug Administration) for the treatment of some lung, skin, kidney, and blood cancers.

The purpose of this study is to find out if treatment with NEO-PV-01 + adjuvant in combination with nivolumab is safe and effective for patients with melanoma, lung, or bladder cancer. The study also will see if NEO-PV-01 vaccine + adjuvant with nivolumab can improve responses compared to available therapies such as nivolumab monotherapy The side effects of NEO-PV-01 + adjuvant and nivolumab will be monitored and additional research tests will be done to assess the immune response against each individual's cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent.
* Have histologically confirmed unresectable or metastatic melanoma having received no more than one prior systemic therapy for the metastatic disease (eg. ipilumamab and/or BRAF inhibitor); unresectable or metastatic smoking-associated NSCLC having received no more than one prior systemic therapy for the metastatic disease (eg standard of care chemotherapy, as appropriate); unresectable or metastatic transitional cell carcinoma of the bladder, urethra, ureter or renal pelvis having received no more than one prior systemic therapy for the metastatic disease.
* Have at least one site of disease measurable disease by RECIST v1.1 that has not been treated with local therapy within 6 months of study treatment. This can be the site for initial or repeat biopsies as long as it will remain measurable following biopsy.
* At least one site of disease must be accessible to provide repeat biopsies for tumor tissue for sequence and immunological analysis.
* Have ECOG PS of 0 or 1 with an anticipated life expectancy of > 6 months.
* Age ≥ 18 years.
* Recovered from all toxicities associated with prior treatment to acceptable baseline status (for laboratory toxicity see below limits for inclusion) or National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03, Grade of 0 or 1, except for toxicities not considered a safety risk (e.g., alopecia or vitiligo).
* Screening laboratory values must meet the following criteria and should be obtained within 30 days (45 if biopsy is repeated) prior to study treatment:
* White blood cell (WBC) count ≥ 3 × 10e3/µL
* Absolute neutrophil count (ANC) ≥ 1.5 × 10e3/µL
* Absolute lymphocyte count (ALC) ≥ 1 × 10e3/µL
* Platelet count ≥ 100 × 10e3/µL
* Hemoglobin > 9 g/dL
* Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 40 mL/min/1.73 m
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN
* Total bilirubin ≤ 1.5 × ULN (except in patients with Gilbert Syndrome who can have total bilirubin < 3.0 mg/dL).
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 7 days prior to the start of nivolumab.
* Female participants, who are not free from menses for >2 years, post hysterectomy / oophorectomy, or surgically sterilized, must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy or to abstain from sexual activity throughout the study, from screening through 5 months after the last dose of study treatment (including nivolumab single agent). Approved contraceptive methods include, for example: intrauterine device, diaphragm with spermicide, cervical cap with spermicide, male condom with spermicide, or female condom with spermicide. Spermicides alone are not an acceptable method of contraception.
* Men who are sexually active with women of child bearing potential must agree to use a condom from screening through 7 months after the last dose of study treatment (including nivolumab single agent).
* For NSCLC, patients must have a minimum of a 10 pack-year smoking history.

Exclusion Criteria:

* Received therapy with any immunotherapeutic agents including, but not limited to, any anti-PD1 or anti-PDL1 antibody therapy, with these exceptions: Melanoma patients having received and progressed on anti-CTLA4 (cyctotoxic T lymphocyte-associated antigen 4) may participate in the trial; Bladder cancer patients having received intra-vesical BCG may participate in the trial.
* Received systemic anti-cancer therapy within 30 days of Week 0, Day 11 of study treatment.
* Have untreated central nervous system (CNS) metastases. Patients are eligible for study participation if CNS metastases are adequately treated and patients are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 60 days prior to consent. In addition, patients must either be off corticosteroids, or on a stable or decreasing dose of 10 mg daily prednisone (or equivalent) for at least 60 days prior to consent.
* Received non-oncology vaccine therapy for prevention of infectious diseases during the 4-week period prior to first dose of nivolumab therapy. Patients may not receive any non-oncology vaccine therapy during the period of NEO-PV-01 + adjuvant or nivolumab administration and until at least 8 weeks after the last dose of the booster vaccine. Annual influenza vaccines are allowed during screening and pre-treatment but not during nivolumab or NEO-PV-01 + adjuvant dosing.
* Received radiation therapy within 4 weeks prior to Week 0, Day 1 of study treatment. Patients may not receive or have received any radiation therapy at the biopsy sites.
* Have an active or history of autoimmune disease (known or suspected). Exceptions are permitted for vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition requiring only hormone replacement, psoriasis not on systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 15 days prior to the first dose of study treatment (nivolumab). Inhaled or topical steroids and adrenal replacement doses (≤ 10 mg daily prednisone equivalents) are permitted in the absence of active autoimmune disease.
* Known human immunodeficiency virus (HIV) infection, active chronic hepatitis B or C, or life-threatening illnesses unrelated to cancer.
* Have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring treatment, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Have any underlying medical condition, psychiatric condition, or social situation that, in the opinion of the Investigator, would compromise study administration as per protocol or compromise the assessment of AEs.
* Have a planned major surgery.
* Pregnant women are excluded from this study because nivolumab, personalized neoantigen peptides, and Poly-ICLC are agents with unknown risks to the developing fetus.
* Nursing women are excluded from this study because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with nivolumab, personalized neoantigen peptides, and Poly-ICLC.
* Have a history of an invasive metastatic disease, except for the following circumstances: individuals with a history of invasive metastatic disease are eligible if they have been disease-free for at least 2 years and are deemed by the Investigator to be at low risk for recurrence of that metastatic disease; individuals with the following cancers are eligible if diagnosed and treated: carcinoma in situ of the breast, oral cavity or cervix, localized prostate cancer, basal cell or squamous cell carcinoma of the skin.
* Mucosal melanoma and uvueal melanoma.
* Patients with NSCLC and known anaplastic lymphoma kinase (ALK) translocations or epidermal growth factor receptor (EGFR) mutations who have not received prior treatment with ALK or EGFR inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events including SAEs and AEs leading to treatment discontinuation | Baseline through 100 days after last dose of nivolumab
  Rate of adverse events including SAEs and AEs leading to treatment discontinuation
Rate of adverse events including SAEs and AEs leading to changes in safety laboratory evaluations | Baseline through 100 days after last dose of nivolumab
  Rate of adverse events including SAEs and AEs leading to changes in safety laboratory evaluations
Rate of adverse events including SAEs and AEs leading to physical examination findings | Baseline through 100 days after last dose of nivolumab
  Rate of adverse events including SAEs and AEs leading to physical examination findings
Rate of adverse events including SAEs and AEs leading to vital signs findings | Baseline through 100 days after last dose of nivolumab
  Rate of adverse events including SAEs and AEs leading to vital signs findings
Rate of adverse events including SAEs and AEs leading to changes in ECOG status | Baseline through 100 days after last dose of nivolumab
  Rate of adverse events including SAEs and AEs leading to changes in ECOG status

SECONDARY OUTCOMES:
Objective response rate (ORR) | Baseline through 104 weeks
  Objective response rate (ORR), defined as the proportion of patients who achieve complete response (CR) or partial response (PR) based on Response Criteria in Solid Tumors (RECIST) v1.1.
Duration of response (DOR) | Baseline through 104 weeks
  Duration of response (DOR), defined as the date of the first documentation of a confirmed response to the date of the first documented PD.
Clinical benefit rate (CBR) | Baseline through 104 weeks
  Clinical benefit rate (CBR), defined as the proportion of patients who achieve CR, PR, or stable disease (SD) based on RECIST v1.1
Response conversion rate (RCR) | Baseline through 104 weeks
  Response conversion rate (RCR) of NEO-PV-01 + adjuvant with nivolumab at Week 24 defined as the proportion of patients who improve in RECIST v1.1 category from Week 12 to Week 24 (e.g., PD to SD/PR/CR, SD to PR/CR, PR to CR).
Progression-free survival (PFS) | Baseline through 104 weeks
  Progression-free survival (PFS), defined as the time from the date of first dosing to the date of first documented PD or death.
Overall survival (OS) | Baseline through 104 weeks
  Overall survival (OS), defined from the date of enrollment and death from any cause.

OTHER OUTCOMES:
Immune Responses | Day 1 of nivolumab through 104 weeks
  Antigen-specificity in peripheral CD8+ and CD4+ T cell responses and tumor biopsies following treatment with NEO-PV-01 + adjuvant and nivolumab

CONTACTS AND LOCATIONS:
Overall Officials: Mark DeMario, MD, Study Director — BioNTech US Inc.
Locations (9):
- United States (9):
  - City of Hope, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poran A, Scherer J, Bushway ME, Besada R, Balogh KN, Wanamaker A, Williams RG, Prabhakara J, Ott PA, Hu-Lieskovan S, Khondker ZS, Gaynor RB, Rooney MS, Srinivasan L. Combined TCR Repertoire Profiles and Blood Cell Phenotypes Predict Melanoma Patient Response to Personalized Neoantigen Therapy plus Anti-PD-1. Cell Rep Med. 2020 Nov 17;1(8):100141. doi: 10.1016/j.xcrm.2020.100141. eCollection 2020 Nov 17. PMID 33294862
- [Derived] Ott PA, Hu-Lieskovan S, Chmielowski B, Govindan R, Naing A, Bhardwaj N, Margolin K, Awad MM, Hellmann MD, Lin JJ, Friedlander T, Bushway ME, Balogh KN, Sciuto TE, Kohler V, Turnbull SJ, Besada R, Curran RR, Trapp B, Scherer J, Poran A, Harjanto D, Barthelme D, Ting YS, Dong JZ, Ware Y, Huang Y, Huang Z, Wanamaker A, Cleary LD, Moles MA, Manson K, Greshock J, Khondker ZS, Fritsch E, Rooney MS, DeMario M, Gaynor RB, Srinivasan L. A Phase Ib Trial of Personalized Neoantigen Therapy Plus Anti-PD-1 in Patients with Advanced Melanoma, Non-small Cell Lung Cancer, or Bladder Cancer. Cell. 2020 Oct 15;183(2):347-362.e24. doi: 10.1016/j.cell.2020.08.053. PMID 33064988